CLINICAL TRIAL: NCT00251225
Title: A Phase II Study of Imatinib and Docetaxel in Metastatic Hormone Refractory Prostate Cancer
Brief Title: A Study of Imatinib and Docetaxel in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leonard Appleman (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Leonard Appleman, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-019
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer
Keywords: prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Imatinib Mesylate; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hormone Refractory Prostate Cancer (Experimental): Gleevec + Docetaxel: Daily Oral Gleevec in Combination with Every-Three-Week Intravenous Docetaxel
  Interventions: Drug: Gleevec; Drug: Docetaxel

INTERVENTIONS:
Drug: Gleevec — Imatinib-400mg po qd for 10 days to commence on day 3. On day 0, Docetaxel 60mg/m^2 administered IV
  Other Names: Imatinib; Imatinib Mesylate; ST1571
Drug: Docetaxel — 60 mg/m^2 administered IV on day 0
  Other Names: Taxotere

SUMMARY:
The purpose of this study is to determine the effectiveness of two drugs, docetaxel and Gleevec®(also called imatinib), in prostate cancer that no longer responds to hormone therapy. The investigators are interested in finding out if the combination of these two drugs is more effective than docetaxel alone in the treatment of prostate cancer.

DETAILED DESCRIPTION:
This is a non-randomized multicenter Phase II trial of Gleevec and docetaxel in chemo naïve metastatic hormone refractory prostate cancer. The primary objective of this study is to assess the time to disease progression in patients with hormone refractory prostate cancer treated with daily oral imatinib and intravenous docetaxel, administered every three weeks. Secondary objectives include: 1) to assess the rate of response to imatinib and docetaxel, using Prostate Specific Antigen (PSA) and/or measurable disease; 2) to assess the overall survival of patients with hormone refractory prostate cancer treated with imatinib and docetaxel; and 3) to evaluate the qualitative and quantitative toxicities of this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a histologic diagnosis of adenocarcinoma of the prostate Stage D2 that is unresponsive or refractory to hormone therapy. Must have metastatic prostate cancer with a rising PSA, and deemed to be hormone refractory.
2. All subjects must have pre-study PSA within 28 days prior to registration
3. Subjects who have measurable disease must have had X-rays, scans or physical examinations used for tumor measurement completed within 28 days prior to registration. Subjects must have non-measurable disease assessed within 28 days (for PSA level) or 42 days (for imaging studies) prior to registration.
4. Subjects with bone metastases, as documented by X-ray, bone scan, MRI, or biopsy.
5. All subjects must have had a CT scan of the abdomen and pelvis within 28 days prior to registration.
6. Subjects must have been surgically or medically castrated. If the method of castration was LHRH (Luteinizing Hormone-Releasing Hormone) agonists, then the subject must be willing to continue the use of LHRH agonists.
7. If the subject has been treated with non-steroidal anti-androgens or other hormonal treatment these agents must have been stopped at least 28 days prior to enrollment for flutamide or ketoconazole, and at least 42 days prior to enrollment for bicalutamide or nilutamide; and the subjects must have demonstrated progression of disease since the agents were suspended.
8. Prior radiation therapy is allowed. At least 21 days must have elapsed since the completion of radiation therapy, and the subject must have recovered from the side effects of the radiation
9. 9. Due to the unknown side effects of imatinib, men of reproductive potential must agree to use an effective contraceptive method.
10. Subjects must have recovered from major infections and/or surgical procedures and, in the opinion of the investigator, not have significant active concurrent other medical illness precluding protocol treatment.
11. ECOG performance status of 0-1
12. ANC ≥ 1,500/mL and a platelet count of ³ 100,000/mL. These tests must be obtained within 7 days prior to registration.
13. Serum bilirubin ≤ 1.3, SGOT and SGPT ≤ 2 x institutional upper limit of normal, and a serum creatinine ≤ 1.8 mg/dl. These tests must be obtained within 7 days prior to registration. Testosterone level may be done 28 days prior to study entry. Testosterone level should be below 50 ng/dL.

Exclusion Criteria:

1. No prior chemotherapy for hormone-refractory disease is allowed. At least three weeks must have elapsed since the completion of any non-cytotoxic investigational therapy, and the patient must have recovered from the side effects of the therapy.
2. No other cytotoxics, biological response modifiers, radiation therapy, corticosteroid or hormonal concomitant therapy (other than continuing LHRH treatment) may be given during protocol treatment. Bisphosphonates may be given during protocol treatment. No unconventional therapy may be given during protocol treatment.
3. Subjects must NOT have Grade III/IV cardiac problems as defined by the New York Heart Association Criteria.
4. Subjects with known chronic liver disease are NOT eligible
5. Must NOT have a known diagnosis of human immunodeficiency virus (HIV) infection.
6. Subjects must NOT have known brain metastases.
7. No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ carcinoma of any site, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-08; Primary Completion 2009-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard J Appleman, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hormone Refractory Prostate Cancer Patients: Patients with hormone refractory prostate cancer treated with Docetaxel 60 mg/m^2 IV every 21 days + Imatinib 400 mg PO daily, or, for 10/21 days
Period: Overall Study
Arm/Group | Hormone Refractory Prostate Cancer Patients
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hormone Refractory Prostate Cancer Patients: Docetaxel 60 mg/m^2 IV every 21 days + Imatinib 400 mg PO daily, or, for 10/21 days
Arm/Group | Hormone Refractory Prostate Cancer Patients
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 69 [54 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Overall Time To Progression (TTP)
Description: TTP is the amount of time from date of registration to date of first documentation of progression or symptomatic deterioration. For progression, one or more of the following must occur: (1) 20% increase in the sum of longest diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline. (2) Increase in PSA by at least 25% from baseline in patients whose PSA did not decrease, and of 50% from nadir in patients whose PSA decreased with a confirmation 3 weeks later. (3) Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). (4) Appearance of any new lesion/site. (5) Death due to disease without prior documentation of progression and without symptomatic deterioration, which is defined as global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: Up to 24 months
Population: Patients with hormone refractory prostate cancer who received at least 1 cycle of Docetaxel + Imatinib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Hormone Refractory Prostate Cancer Patients
Number analyzed (Participants) | 29
months | 6.4 [4.8 to 8.4]

2. Secondary Outcome: Prostate-Specific Antigen (PSA) Response Rate
Description: PSA response rate is the number of participants who experienced a best response of: complete response, CR (PSA less than or equal to 0.2 ng/mL, documented two or more times, a minimum of four weeks apart), partial response, PR (a decline in PSA by at least 50%, confirmed by a second PSA value four or more weeks later) or stable disease (does not qualify for CR, PR, Progression or Symptomatic Deterioration, at least 6 weeks after registration) / total number of analyzable patients.
Time Frame: Up to 12 months
Population: Patients with hormone refractory prostate cancer who received at least 1 cycle of Docetaxel + Imatinib
Measure: Number; unit: percentage of patients
Arm/Group | Hormone Refractory Prostate Cancer Patients
Number analyzed (Participants) | 29
percentage of patients | 72.4

3. Secondary Outcome: Overall Survival (OS)
Description: OS is the amount of time in months from the date of registration to the date of death from any cause.
Time Frame: Up to 60 months
Population: Patients with hormone refractory prostate cancer who received at least 1 cycle of Docetaxel + Imatinib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Hormone Refractory Prostate Cancer Patients
Number analyzed (Participants) | 29
months | 23.1 [11.5 to 34.7]

ADVERSE EVENTS:
Arm/Group | Hormone Refractory Prostate Cancer Patients
Serious Adverse Events (participants affected / at risk) | 35/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hormone Refractory Prostate Cancer Patients (N=49)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Alkaline phosphatase (Investigations) | 1
Calcium, serum-low (hypocalcemia) (Investigations) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Cardiovascular/Arrhythmia-Other (Cardiac disorders) | 1
Cardiovascular/General-Other (Cardiac disorders) | 1
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 1
Heartburn/dyspepsia (General disorders) | 1
Hematochezia (General disorders) | 1
Hemorrhage, GI, Duodenum (Vascular disorders) | 1
Hemorrhage, GI, Upper GI NOS (Vascular disorders) | 1
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 1
Hemorrhage-Other (Vascular disorders) | 1
Hypocalcemia (Investigations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection - Other (Specify, __) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Lung (pneumonia) (Infections and infestations) | 1
Infection/Febrile Neutropenia-Other (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Obstruction, GU, Ureter (Renal and urinary disorders) | 1
Secondary Malignancy-Other (excludes metastasis from initial primary) (General disorders) | 1
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Ventricular arrhythmia, Ventricular fibrillation (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 3
Febrile neutropenia (fever of unknown origin)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Infections and infestations) | 4
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 11
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hormone Refractory Prostate Cancer Patients (N=49)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 14
Hemoglobin (Blood and lymphatic system disorders) | 17
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 17
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia, Atrial flutter (Cardiac disorders) | 1
Ventricular arrhythmia, PVCs (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia, Sinus tachycardia (Cardiac disorders) | 3
Left ventricular diastolic dysfunction (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 3
Hypotension (Cardiac disorders) | 3
Constitutional Symptoms - Other (Specify, __) (General disorders) | 2
Sweating (diaphoresis) (General disorders) | 2
Weight loss (General disorders) | 3
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 4
Rigors/chills (General disorders) | 4
Insomnia (General disorders) | 7
Fatigue (asthenia, lethargy, malaise) (General disorders) | 35
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3
Flushing (Skin and subcutaneous tissue disorders) | 3
Nail changes (Skin and subcutaneous tissue disorders) | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 10
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 4
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 7
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 7
Dehydration (Gastrointestinal disorders) | 9
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 13
Anorexia (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 24
Hemorrhage, GI, Lower GI NOS (Vascular disorders) | 2
Hemorrhage, GI, Rectum (Vascular disorders) | 2
Infection (documented)w Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) Liver (Infections and infestations) | 1
Infection (documented) w Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L), Urinary tract NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Upper airway NOS (Infections and infestations) | 1
Infection with unknown ANC, Upper airway NOS (Infections and infestations) | 1
Infection - Other (Specify, __) (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils, Urinary tract NOS (Infections and infestations) | 3
Lymphatics - Other (Specify, __) (Blood and lymphatic system disorders) | 1
Edema: head and neck (Blood and lymphatic system disorders) | 4
Edema: limb (Blood and lymphatic system disorders) | 12
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Glucose, serum-low (hypoglycemia) (Investigations) | 1
Calcium, serum-low (hypocalcemia) (Investigations) | 2
Potassium, serum-low (hypokalemia) (Investigations) | 3
Alkaline phosphatase (Investigations) | 4
Glucose, serum-high (hyperglycemia) (Investigations) | 6
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Whole body/generalized (Musculoskeletal and connective tissue disorders) | 3
Confusion (Nervous system disorders) | 1
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1
Mood alteration, Depression (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Neurology - Other (Specify, __) (Nervous system disorders) | 7
Neuropathy: sensory (Nervous system disorders) | 11
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1
Vision-flashing lights/floaters (Eye disorders) | 1
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2
Watery eye (epiphora, tearing) (Eye disorders) | 2
Pain, Neck (General disorders) | 1
Pain - Other (Specify, __) (General disorders) | 2
Pain, Abdomen NOS (General disorders) | 2
Pain, Joint (General disorders) | 2
Pain, Chest/thorax NOS (General disorders) | 3
Pain, Muscle (General disorders) | 3
Pain, Bone (General disorders) | 4
Pain, Head/headache (General disorders) | 4
Pain, Extremity-limb (General disorders) | 5
Pain, Back (General disorders) | 9
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Urine color change (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes